CLINICAL TRIAL: NCT06310863
Title: Pivotal Study to Evaluate the Efficacy and Safety of Injection With LASBEAU Strong as Compared to Restylane® Lyft Lidocaine in Temporary Correction of Nasolabial Folds
Brief Title: Pivotal Study to Evaluate the Efficacy and Safety of Injection With LASBEAU Strong in Correction of Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Chong Hyun Won, professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EXOCOBIO-NASAL-01
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Dermal Fillers
Keywords: LASBEAU Strong; hyaluronic acid; lidocaine; nasolabial fold

STUDY DESIGN:
Intervention Model Description: Randomized, Matched pairs, Active controlled
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): The test device, LASBEAU Strong, was developed for the purpose of temporary improvement of facial nose and lip wrinkles, which is the same indication as the control device, and has a hyaluronic acid structure similar to that of Restylane® Lyft Lidocaine, and was developed using the same crosslinker, 1,4-butanediol diglycidyl ether. The test device, LASBEAU Strong, has a higher content of hyaluronic acid than the control device, Restylane® Lyft Lidocaine, but the clinical efficacy cannot be evaluated as superior because of the high content of hyaluronic acid. This is because, in addition to the content of hyaluronic acid, differences in the manufacturing process can affect the physicochemical properties and decomposition period.
  Interventions: Device: LASBEAU Strong or Restylane Lyft injection as hyaluronic acid fillers
- control group (Active Comparator): Restylane® Lyft Lidocaine, a previously licensed product with the same ingredients as the test group, was selected as the control group. Restylane® Lyft Lidocaine is a representative filler formulation that has been recognized for the temporary improvement of facial nose and lip wrinkles, and it was selected as a control group because it is similar to the clinical trial medical device in the test group, and the application site and application method are the same. The control device, Restylane® Lyft Lidocaine, is a product imported and sold by Galderma Korea, which is a bacterial fermentation product and is known as non-animal hyaluronic acid. The purpose of use is to temporarily improve the wrinkles of the nose and lips of the face.
  Interventions: Device: LASBEAU Strong or Restylane Lyft injection as hyaluronic acid fillers

INTERVENTIONS:
Device: LASBEAU Strong or Restylane Lyft injection as hyaluronic acid fillers — Subjects will be randomized to receive LASBEAU Strong or Restylane Lyft injections into each of the nasolabial folds on both sides.
  LASBEAU Strong or Restylane Lyft Injection Box

SUMMARY:
Background: Nonsurgical injectable treatments have become popular for aesthetic purposes. In recent years, cross-linked hyaluronic acid (HA) fillers containing lidocaine have been used to correct the nasolabial folds.

Aim: The aim of this study was to demonstrate the efficacy and safety of a new HA filler (LASBEAU Strong) (24 mg/mL) compared with a conventional HA filler (Restylane Lyft) for the restoration of nasolabial folds.

Patients/methods: A total of 72 subjects were enrolled and randomized to receive injections of the new HA filler (test group) or the conventional HA filler (control group) on the left or right side of the face. The mean value difference in the Wrinkle Severity Rating Scale (WSRS) scores at week 24 evaluated primary efficacy. The WSRS and the Global Aesthetic Improvement Scale (GAIS) at weeks 8, 16, 24, and 48 evaluated secondary efficacy. Adverse events, laboratory tests, and a check of vital signs at every visit assessed safety.

DETAILED DESCRIPTION:
1. Introduction

   Hyaluronic acid (HA) is a type of glycosaminoglycan that has a repeating structure of sodium glucuronate and N-acetylglucosamine unit sugar and that is known as a component of connective tissue such as joint fluid, oculovitreous fluid, umbilical cord, dermis surface layer, etc. The main function of HA in the extracellular matrix is to stabilize the extracellular structure and form matrix fluid. HA has strong hydrophilicity and functions as a natural supply of moisture to the skin, contributing to its flexibility and swelling. In view of its structural role in tissues, protective effect on cell membranes, and viscoelasticity, HA is ideal as a skin filler. Cross-linking is a process in which HA in a liquid state is transformed into a soft solid or gel by chemically combining each chain of HA. By slowing down HA metabolism in the human body, cross-linked HA can have a long-lasting effect in terms of beauty. Among nonsurgical procedures for wrinkle improvement, soft tissue augmentation using an injectable filler is one of the most frequently performed cosmetic procedures and is widely applied. However, there has been a risk of a serious hypersensitivity reaction due to an immune response caused by various substances. Among them, since HA is a form of polymer with the same structure in all species, cross-linked and nonanimal-stabilized HA derivatives have longer-lasting power and less immune response. The new HA filler is a biomaterial that contains nonanimal-stabilized HA derived from bacterial fermentation and lidocaine, a local anesthetic that reduces pain during the procedure. This product is a cross-linked HA gel, a biomaterial for tissue repair, and was developed to temporarily improve facial wrinkles in the adult face and relieve pain during the procedure. The aim of this trial was to demonstrate that the new HA filler consisting of 24 mg/mL cross-linked HA containing lidocaine was not inferior to the conventional HA filler, which contains the same ingredient for the temporary restoration of nasolabial folds with moderate to severe Wrinkle Severity Rating Scale (WSRS) scores.
2. Materials and methods

2.1 Trial design

This multicenter, randomized, double-blind, split-face clinical trial was conducted from November 2019 to February 2021 at two investigational sites (Asan Medical Center and Nowon Eulji Medical Center) in the Republic of Korea. This trial protocol was approved by the institutional review board of both institutions and followed the guidelines of the 1975 Declaration of Helsinki. All subjects provided written informed consent, including a signed photographic consent form, before participation in the trial.

2.2 Trial population

From November 2019 to June 2020, among subjects who desired temporary improvement of the nasolabial folds on both sides, those who had a WSRS of 3 or 4 points (they didn't must have the same score on both sides) were enrolled in the trial. Subjects aged over 19 years were included in the trial. The subjects agreed not to have any other treatment for facial wrinkle correction during the trial period. The exclusion criteria were administration of antithrombotic agents (excluding low-dose aspirin therapy: 100 mg; maximum 300 mg/day) from 2 weeks before to 2 weeks after the injection of the HA fillers; administration of vitamin E preparations or NSAID preparations from 1 week before to 1 week after the injection of the HA fillers; previous or current bleeding disorders; calcium hydroxyapatite (CaHA) or poly L-lactide (PLLA) filler treatment within 1 year after the screening date; use of topical agents (steroids or retinoids: only for pharmaceuticals, excluding cosmetics) on the face within 4 weeks after the screening date or planning to use them during the clinical trial period (however, for treatment purposes, steroid ointments could be used for a short period within 14 consecutive days); administration of antiwrinkle therapy, acne scar treatment, plastic surgery (including botulinum toxin injection), facial abrasion, or skin rejuvenation within the past 24 weeks; permanent skin expansion implant, such as soft form and silicon on the face; skin disorders; wound infections on the face; and a history of keloid or hypertrophic scar. Other exclusion criteria were disagreement to contraception by a medically allowed method for the trial period after the injection of the HA fillers among female subjects who were probably pregnant; pregnancy or lactation; and clinically significant findings considered inappropriate for this test by the investigator.

2.3 Materials

LASBEAU Strong (ExocoBio, Inc., Seoul, Korea), an investigational device filled with a colorless transparent liquid filler consisting of 24 mg/mL cross-linked HA containing lidocaine, was used as a test device in the trial.

Restylane Lyft (GalDerma a Korea, Inc., Seoul, Korea), a filler filled with cross-linked HA containing lidocaine, was used as a control device.

2.4 Trial protocol

At the treatment visit (week 0), the subjects were randomized to determine into which nasolabial fold the test filler would be injected; the control filler was injected into the other nasolabial fold. After the HA filler injections, the subject was kept under observation for 30 min to check for adverse events (AEs). The subjects received a subject diary and recorded the occurrence and disappearance of AEs in the subject diary for 2 weeks; the subjects returned the subject diary at week 8. The response to the injection of the test and control fillers was documented at weeks 8, 16, and 24. The call visit at week 36 performed additional safety assessment. At week 48, the subjects completed the trial, and evaluated the safety and efficacy of the treatment.

2.5 Treatment procedure

Before the HA filler injections, the treatment site was cleansed with disinfecting fluid. Subjects were applied to the test filler to one side of the face and the control filler to the contralateral side. Following the injection of the two fillers, the injection sites were massaged as needed.

2.6 Methods of randomization and blinding

A random-number table was used for randomization. The investigator opened the randomization envelopes in the order in which the subjects were registered and injected each HA filler. To maintain blindfolding between the subjects and the independent investigators until the end of the trial, the subjects and the independent investigators did not know into which side of the nasolabial fold the test filler and the control filler were injected. The investigator opened the randomization envelope immediately before the HA filler injections, so that the investigator knew the fillers to be injected for each nasolabial fold. Before the HA filler injections and at each follow-up visit, high-quality digital photographs, including the left and right nasolabial folds, were taken. It was necessary to ensure that the left and right sides were symmetrical from the beginning of the nose lip fold to the tip of the chin, centering on the center line of the lips. Any information about the subjects was removed from the photographs, which were then sent to independent investigators to assess the efficacy of the treatment.

2.7 Efficacy assessment

The primary efficacy measure was mean value differences in the WSRS scores assessed by three independent investigators between baseline and 24 weeks (Table 1). WSRS scores were first evaluated by the independent investigators. If the WSRS scores were the same among independent investigators, they were accepted. If the WSRS scores were different, they were evaluated by different independent investigators, and results of the same values were adopted and interpreted. The difference in the mean values of WSRS scores between the test group and the control group was then calculated.

The investigators evaluated WSRS and GAIS (Global Aesthetic Improvement Scale) scores at each follow-up visit as secondary endpoints. The independent investigators evaluated the proportion of subjects with an improvement in WSRS scores of one or more points at weeks 24 and 48. The subjects' pretreatment photographs served as reference images for assessing improvement. Additional visits were performed at weeks 36 (call visit) and 48 following the HA filler injections. At week 36, a call visit was made to check for AEs and concomitant medications; at week 48, the subjects visited the hospital, took photography of the injection sites and WSRS or GAIS evaluation were performed.

2.8 Safety assessment

Adverse events (AEs) and serious adverse events (SAEs) that occurred following the HA filler injections were presented as numbers of subjects, percentages, and incidences.

2.9 Statistical analyses

The primary efficacy endpoint was the mean value difference in WSRS scores between the test group and the control group, as determined by the independent investigators at week 24.

The secondary efficacy endpoints included the following: (1) The investigators calculated the mean value differences in the WSRS scores between the test group and the control group at weeks 8, 16, 24, and 48 after the filler injections. (2) The investigators calculated the mean value differences in the GAIS scores between the test group and the control group at weeks 8, 16, 24, and 48 after the filler injections. (3) The independent investigators calculated whether the ratio of subjects whose WSRS scores improved by one or more points in the test group and the control group compared with those before the filler injections at weeks 24 and 48. The two-sample t-test and Wilcoxon's rank sum test were used for the analyses of endpoints (1) and (2). The chi-square test and Fisher's exact test were used for the analysis of endpoints (3). The chi-square test and Fisher's exact test were used for the safety analysis. The comparisons were subjected to two-tailed tests with a 5% significance level. The paired t-test, Wilcoxon's signed rank test and McNemar's test analyzed the laboratory test results, vital signs, and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

- 1. Men and women over 19 years of age 2. Subjects who wish to temporarily improve their nasolabial folds, those who have a Wrinkle Severity Rating Scale (WSRS) of 3 or 4 points (both do not have to have the same score) 3. Subjects who agree to discontinue all dermatological treatments or treatments (filler, botulinum toxin, laser treatment, chemical exfoliation, cosmetic surgery, etc.) other than the application of clinical trial medical devices during this clinical trial period 4. Can understand and follow instructions, and participate in the pre-clinical period.

5. Subjects who voluntarily decide to participate in this clinical trial and agree in writing to the informed consent form.

Exclusion Criteria:

* 1. Subjects who administered anti-thrombotic agents (excluding low-dose aspirin (100 mg, up to 300 mg/day) from 2 weeks to 2 weeks after clinical trial application), Vitamin E formulation, and NSAID formulation from 1 week to 1 week after application 2. Subjects with a history of bleeding at the past or present time 3. Subjects who received CaHA (Calcium Hydroxyapatite) or Poly L-Lactide (PLA) filler treatment at the site where the clinical trial device is applied within one year from the screening date 4. Subjects who used local application agents (steroids, retinoids: medicines only) on their face within 4 weeks from the screening date or who are scheduled to use them during the clinical trial (but steroid ointment can be used for a short period of 14 consecutive days for treatment purposes) 5. Subjects who used immunosuppressants, chemotherapy drugs, or systemic corticosteroids within 12 weeks from the screening date 6. Subjectswho received treatment for wrinkle improvement or acne scars within 24 weeks from the screening date 7. Subjects who underwent skin peeling, skin regeneration, or plastic surgery (including botulinum toxin injection) on their face within 24 weeks from the screening date 8. Subjects with the permanent skin-expanding prosthesis such as a cured gel or silicone into the face 9. Subjects with a skin disease or wound infection in the face that affects this clinical trial 10. Those with an autoimmune disease or a history of it or a weakened immune system 11. Those with a history of symptoms of anaphylaxis or severe complex allergies 12. Those with a history of hypertrophic scarring or keloidosis 13. Patients with hypersensitivity to lidocaine or other amide-based local anesthetics 14. A person who has or currently has a severe clinical impairment in the cardiovascular system, digestive system, respiratory system, endocrine system and central nervous system, or has a mental illness that significantly affects this clinical trial 15. Those who participated in other clinical trials within 30 days from the date of screening and received/applied clinical trial medicines/clinical medical devices 16. Among female subjects who are likely to become pregnant, those who do not agree to use contraception* in a medically permitted manner up to 48 weeks after the application of the clinical trial medical device

  * Medically permitted contraception methods: condoms, oral contraception lasting at least three months, using contraceptives for injection or insertion, and installing intrauterine contraceptive devices, etc.

    17. Pregnant or lactating woman 18. Anyone who has any clinical significance findings deemed inappropriate for this test by the person in charge or in charge of the test as medically determined above

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Differences in the mean value of the Wrinkle Severity Rating Scale (WSRS) between the test group and the control group | at 24 weeks after the application of the clinical trial medical device
  Differences in the mean value of the Wrinkle Severity Rating Scale (WSRS) between the test group and the control group evaluated by independent investigators

SECONDARY OUTCOMES:
The mean value differences in the WSRS scores between the test group and the control group | at weeks 8, 16, 24, and 48 after the filler injections
  The investigators calculated the mean value differences in the WSRS scores between the test group and the control group
Differences in GAIS mean values between test and control groups | at weeks 8, 16, 24, and 48 after the filler injections
  The investigators calculated the mean value differences in the GAIS scores between the test group and the control group
Percentage of subjects with WSRS score improvement of at least 1 point | at 24 and 48 weeks after medical device application
  The independent investigators calculated whether the ratio of subjects whose WSRS scores improved by one or more points in the test group and the control group compared with those before the filler injections

CONTACTS AND LOCATIONS:
Overall Officials: Chong Hyun Won, Doctor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan mediccal center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho JY, Kim SH, Cho H, Park Y, Yang HJ, An JS, Won CH, Lee JH. Noninferiority Study Comparing the Efficacy and Safety of a New Hyaluronic Acid (HA) Filler Containing Lidocaine With an Existing HA Filler for the Treatment of Nasolabial Fold Wrinkles: A Randomized, Double-Blind, Split-Face Trial. J Cosmet Dermatol. 2025 Jul;24(7):e70309. doi: 10.1111/jocd.70309. PMID 40620129